CLINICAL TRIAL: NCT03592862
Title: A Randomized, Double-blind, Placebo Controlled, Dose Ranging Study to Assess the Safety, Tolerability, and Efficacy of HTL0018318 in Patients With Dementia With Lewy Bodies
Brief Title: A Study to Assess Safety, Tolerability, and Efficacy of HTL0018318 in Patients With Dementia With Lewy Bodies
Acronym: DLB
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Pending investigation of an unexpected animal toxicology finding.
Sponsor: Nxera Pharma UK Limited (Industry)
Collaborators: Sosei (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HTL0018318-203
Record Dates: First submitted 2018-06-25; First posted 2018-07-19 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Dementia With Lewy Bodies
MeSH Terms: conditions — Lewy Body Disease

STUDY DESIGN:
Intervention Model Description: Placebo controlled
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HTL0018318 high dose (Experimental): oral capsule, once daily
  Interventions: Drug: HTL0018318
- HTL0018318 mid dose (Experimental): oral capsule, once daily
  Interventions: Drug: HTL0018318
- HTL0018318 low dose (Experimental): oral capsule, once daily
  Interventions: Drug: HTL0018318
- Placebo (Placebo Comparator): oral capsule, once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HTL0018318 — Oral capsule
  Arms: HTL0018318 high dose; HTL0018318 low dose; HTL0018318 mid dose
Drug: Placebo — Oral capsule
  Arms: Placebo

SUMMARY:
To establish the safety and efficacy of HTL0018318 compared with placebo when administered once daily for 12 weeks to patients with dementia with Lewy bodies.

DETAILED DESCRIPTION:
To assess the safety, tolerability and efficacy of HTL0018318 at 3 dose levels (once daily) compared with placebo over a 12-week treatment period in patients with dementia with Lewy bodies (DLB). Approximately 140 DLB patients who have not received donepezil (Aricept®) and/or other acetyl cholinesterase inhibitors (AchEi) and approximately 32 DLB patients who have had prior treatment experience with donepezil but have stopped usage will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with probable DLB according to the fourth revision of consensus diagnostic criteria for DLB.
* Clinical imaging evidence from either SPECT or MIBG cardiac scintigraphy that is consistent with a clinical diagnosis of DLB.
* Partner or caregiver able to support the patient for the duration of the clinical trial.

Exclusion Criteria:

* Patients with a diagnosis of Parkinson disease at least 1 year prior to onset of dementia.
* Patients with the presence of severe extrapyramidal symptoms
* Patients with the presence of an illness/condition apart from DLB that could contribute to cognitive dysfunction
* Patients with poorly controlled hypertension despite lifestyle modifications and/or pharmacotherapy, who are currently on more than 2 different antihypertensive treatments
* Patients with prominent, recurrent episodes of syncope are related to orthostatic hypotension
* Patients with pulmonary disease or evidence of clinically significant moderate or severe pulmonary symptoms
* Patients who are taking a range of prohibited and restricted medication
* Patients who have been prescribed individualised cognitive rehabilitation, stimulation or training that was performed under medical supervision in the 6 months prior to the screening visit
* Patients who have any known condition(s) that may be contraindicated or interfere with the completion of the nuclear imaging scans.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment related adverse events | Baseline to 12 weeks
  Comparison of HTL0018318 treatment with placebo
Change in systolic, diastolic blood pressure and heart rate | Baseline to 12 weeks
  Comparison of HTL0018318 treatment with placebo

SECONDARY OUTCOMES:
Change from baseline in measures of cognitive impairment | Baseline to 12 weeks
  Comparison of HTL0018318 treatment with placebo
Change from baseline in measures of psychosis (i.e. hallucinations and delusions) | Baseline to 12 weeks
  Comparison of HTL0018318 treatment with placebo

CONTACTS AND LOCATIONS:
Overall Officials: Tim Tasker, MBBS, Study Chair — Heptares Therapeutics Ltd.
Locations (3):
- Japan (3):
  - Nishitaga Hospital, Sendai
  - Kagawa Prefectural Central Hospital, Takamatsu
  - Kurumi Clinic, Tokyo

IPD SHARING:
Plan to Share IPD: No